CLINICAL TRIAL: NCT06005896
Title: A Clinical Model to Predict Successful Renal Replacement Therapy (RRT) Discontinuation in Patients With Acute Kidney Injury (AKI)
Brief Title: A Clinical Model for Dialysis Discontinuation in AKI
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 51678521.0.0000.0068
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Acute Renal Failure; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Success: Patients who were alive and free from RRT 7 days after interrupting RRT.
- Failure: Patients who were not alive or who needed to dialyse again after interrupting RRT for at least 48h.

SUMMARY:
A retrospective study evaluating AKI patients in whom RRT was interrupted for at least 48 hours. Patients who were still RRT-independent 7 days after initial RRT cessation were included in the "Success" group, as opposed to the "Failure" group. Baseline characteristics and variables at the time of RRT interruption were collected. Multivariable analysis was performed and a model was generated to evaluate the prediction of success.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving kidney replacement therapy due to AKI from October 2020 to February 2022 were considered for inclusion in the study. Patients who managed to remain at least 48 consecutive hours without receiving kidney replacement therapy prescription were included.

Exclusion Criteria:

* Patients who had kidney replacement therapy interrupted exclusively due to haemodynamic instability, death or decision for palliative care were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients from a large tertiary care hospital receiving kidney replacement therapy due to AKI.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Success in RRT discontinuation | 7 days
  To be alive and free from RRT 7 days after interrupting RRT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo School of Medicine, São Paulo, São Paulo, Brazil